CLINICAL TRIAL: NCT05290545
Title: A Comparative Study of Haploidentical Transplantation Supported by Third-party Cord Blood and Haploidentical Transplantation in Hematological Malignancies
Brief Title: Haplo-PBSC+Cord vs Haplo-PBSC+BM for Hematological Malignancies Undergoing Allo-HSCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Hunan Provincial People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); First People's Hospital of Chenzhou (Other); Dongguan People's Hospital (Other Government); The First People's Hospital of Guangzhou (Unknown)
Responsible Party: Principal Investigator, Liu Qifa, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2021-126
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2022-03

CONDITIONS: Hematological Malignancies; Hematopoietic Stem Cell Transplantation
Keywords: Hematological malignancies; Haploidentical transplantation; Umbilical cord blood; Disease-free survival
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo-PBSC+Cord group (Experimental): The third party UCB will be infused the day after infusion of PBSCs from HID.
  Interventions: Other: PBSCs; Other: Cord
- Haplo-PBSC+BM group (Active Comparator): The BMSCs from the same HID will be infused the day after infusion of PBSCs.
  Interventions: Other: PBSCs; Other: BMSCs

INTERVENTIONS:
Other: PBSCs — PBSCs harvest is performed from day 5 of G-CSF to obtain at least 7.0×10^8 total nucleated cells/kg recipient ideal body weight.
Other: Cord — The criteria for cord selection included the following: (1) ≥3 of 6 HLA loci , (2) blood type matches, (3) contained a minimum cell count of 0.3×10^8 nucleated cells/kg and 0.15×10^6 CD34-positive cells/kg before freezing. The third party UCB will be infused the day after infusion of PBSCs.
  Arms: Haplo-PBSC+Cord group
Other: BMSCs — BMSCs of donor will be collected and infused at least 0.5×10^8 total nucleated cells/kg recipient ideal body weight the day after PBSCs infusion.
  Arms: Haplo-PBSC+BM group

SUMMARY:
The objective of this study was to explore whether the combination with umbilical cord blood (UCB) is associated with superior disease-free survival (DFS) in the setting of haploidentical donors (HID) transplantation.

DETAILED DESCRIPTION:
The main causes of allogeneic hematopoietic stem cell transplantation (allo-HSCT) failure are primary disease relapse and transplant-related complications, especially relapse. In recent years, with the development of transplantation technology, alternative donors such as HID and UCB have been widely used. But, these alternative donors are associated with high incidences of transplant-related complications and mortalities when compared with human leukocyte antigen (HLA)-matched donors. Some studies suggeted that mixed grafts might overcome the disadvantages of a single alternative graft. UCB transplant (UCBT) supported by third-party HID or HID transplants supported by third-party UCB has been reported to have rapid engraftment and low incidences of graft-versus-host-disease (GVHD), making survival improvement. However, most of these results came from single-arm studies. The comparative studies between haplo-PBSC+Cord and haplo-PBSC+BM are scarce in the setting of HID transplantation. In a retrospective study, the investigators found haplo-PBSC+Cord transplantation has superior DFS than haplo-PBSC+BM in hematological malignancies. To further confirmed this conclusion, the investigators plan to conduct a prospective, multicenter, phase 3 randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies undergoing first HID allo-HSCT
* Age 18 to 65 years old with ECOG performance status 0-2
* Received myeloablative conditioning regimens
* Sign informed consent form, have the ability to comply with study and follow-up procedures

Exclusion Criteria:

* Received PBSCs as only grafts
* Acute leukemia transformed from a myeloproliferative tumor
* Cardiac dysfunction (particularly congestive heart failure, unstable coronary artery disease and serious cardiac ventricular arrhythmias requiring antiarrhythmic therapy)
* Respiratory failure ( PaO2 ≤60mmHg)
* Hepatic abnormalities (total bilirubin ≥3 mg/dL, aminotransferase >2 times the upper limit of normal)
* Renal dysfunction (creatinine clearance rate < 30 mL/min)
* ECOG performance status 3, 4 or 5
* With any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 1 year

SECONDARY OUTCOMES:
Relapse rate | 1 year
Overall survival (OS) | 1 year
The cumulative incidence of hematopoietic engraftment. | 30 days post-transplantation
  Hematopoietic engraftment includes the time of neutrophil and platelet engraftment. Neutrophil engraftment was defined as the first of two consecutive days with an absolute neutrophil count in the peripheral blood exceeding 0.5 × 10^9/L and the platelet engraftment was defined as the first of 3 days with an absolute platelet count exceeding 20 × 10^9 /L without transfusion support.
The cumulative incidence of acute graft-versus-host-disease (GVHD) | 100 days post-transplantation
  Acutue GVHD was defined according to the 1994 consensus conference on acute GVHD grading and graded from I to IV.
The cumulative incidence of chronic GVHD | 1 year
  Chronic GVHD was graded as mild, moderate and severe according to the national institutes of health consensus development project on criteria for clinical trials in chronic GVHD: the 2014 diagnosis and staging working group report.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu S, Huang F, Xu N, Zhang Z, Liu C, Xu X, Fan Z, Zeng X, Liu Q, Qiu G, Xi X, Lin R, Liang X, Jiang Y, Dai M, Jin H, Li X, Wang S, Wu M, Sun J, Xuan L, Liu Q. Haploidentical peripheral blood stem cells combined with bone marrow or unrelated cord blood as grafts for haematological malignancies: an open-label, multicentre, randomised, phase 3 trial. Lancet Haematol. 2025 Mar;12(3):e190-e200. doi: 10.1016/S2352-3026(24)00372-7. Epub 2025 Feb 4. PMID 39919775